CLINICAL TRIAL: NCT00036283
Title: Clinical Protocol For A Phase II Double-Blind, Placebo-Controlled, Randomized Study Of Celecoxib (Sc-58635) In Oral Premalignant Lesions, Investigator IND
Brief Title: Chemoprevention of Oral Premalignant Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NQ4-00-02-011
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Precancerous Conditions
MeSH Terms: conditions — Precancerous Conditions | interventions — Celecoxib

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
Reduction in size and number of oral premalignant lesions

ELIGIBILITY:
Inclusion Criteria:

* 8mm oral premalignant lesion that has not been biopsied in the past 6 months

Exclusion Criteria:

* Taking >100mg daily dose of NSAIDS (Non-steroidal anti-inflammatory drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2000-11; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of celecoxib in subjects with Early or Advanced oral premalignant lesion (OPL)
by both clinical response (reduction in size of all lesions,
prevention of growth in the index lesion and of any new lesions)
and histological response (change in histological grade).
To evaluate the safety of chronic multiple dosing of celecoxib in this patient population.

SECONDARY OUTCOMES:
To evaluate the treatment effects in modulating the expression of genomic and proliferative markers after 12 weeks of treatment with study drug, followed by 12 weeks off study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NQ4-00-02-011&StudyName=Chemoprevention+of+Oral+Premalignant+Lesions